CLINICAL TRIAL: NCT04018768
Title: Multimodal Analgesia With NSAID vs. Narcotics Alone After Shoulder Instability Surgery
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-01177
Record Dates: First submitted 2019-05-29; First posted 2019-07-12 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Ibuprofen; Oxycodone; Acetaminophen; oxycodone-acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ibuprofen + Percocet
  Interventions: Other: ibuprofen 600 mg; Other: Oxycodone/acetaminophen (Percocet) 5 mg/325
- Percocet
  Interventions: Other: Oxycodone/acetaminophen (Percocet) 5 mg/325

INTERVENTIONS:
Other: ibuprofen 600 mg — MRN ending in an EVEN # will receive ibuprofen 600 mg to be taken every 8 hours (TID) as needed (PRN) and oxycodone/acetaminophen (Percocet) 5 mg/325 mg for pain that is not adequately controlled by the ibuprofen.
  Groups: Ibuprofen + Percocet
Other: Oxycodone/acetaminophen (Percocet) 5 mg/325 — MRN ending in an ODD #: will receive the current standard of care postoperative pain management, which is Percocet 5 mg/325 mg every 6 hours PRN.

SUMMARY:
This will be a single-center, prospective observational study. The study will compare post- operative pain scores and narcotic consumption between two groups of patients - one cohort will receive ibuprofen (Motrin) and Percocet (to be used as needed) while the other cohort will receive only Percocet. Both pain management options are considered to be standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II
* Patients scheduled for arthroscopic shoulder instability surgery

Exclusion Criteria:

* Contraindication to ibuprofen or oxycodone/acetaminophen (e.g. hypersensitivity, history of GI or bleeding disorder)
* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age or older than 65
* Any patient considered a vulnerable subject
* Patients on pain medication prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for isolated arthroscopic shoulder instability surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Score | 30 Minutes, 1 Hour Post Surgery, 2 Hours Post Surgery, 3 Hours Post Surgery, 4 Hours Post Surgery
  Scale consisting of a drawn line from 0 to 100 - the patient will be asked to mark where they believe their pain is (100 being worse pain).
Change in Verbal Rating Scale (VRS) | 30 Minutes, 1 Hour Post Surgery, 2 Hours Post Surgery, 3 Hours Post Surgery, 4 Hours Post Surgery
  Consisting of 4 points (0 = no pain, 1 = mild, 2 = moderate, and 3 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Campbell, Principal Investigator — New York Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Bloom DA, Baron SL, Luthringer TA, Alaia MJ, Strauss EJ, Jazrawi LM, Campbell KA. Preoperative Opioid Education has No Effect on Opioid Use in Patients Undergoing Arthroscopic Rotator Cuff Repair: A Prospective, Randomized Clinical Trial. J Am Acad Orthop Surg. 2021 Oct 1;29(19):e961-e968. doi: 10.5435/JAAOS-D-20-00594. PMID 33306558